CLINICAL TRIAL: NCT04009369
Title: Impacts of Physiotherapy Services in a Quebec Emergency Department - Randomized Clinical Trial
Brief Title: Impacts of Physiotherapy Services in a Quebec Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rose Gagnon (Other)
Collaborators: CHU de Quebec-Universite Laval (Other); Integrated University Health and Social Services Center of the Capitale-Nationale (Other); Laval University (Other)
Responsible Party: Sponsor-Investigator, Rose Gagnon, Master's Student, Laval University
Organization: Laval University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MP-20-2019-4307
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Musculoskeletal Pain; Musculoskeletal Diseases; Musculoskeletal Injury
Keywords: Health care access; Health services; Professional practices
MeSH Terms: conditions — Musculoskeletal Pain; Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emergency Physician Group (No Intervention): Usual care by the EP without the intervention of the ED PT.
- Physical Therapist Group (Experimental): Direct access to a PT in the ED immediately after triage and prior to physician assessment.
  Interventions: Other: Direct access to a PT

INTERVENTIONS:
Other: Direct access to a PT — Direct access to a PT in the ED immediately after triage and prior to physician assessment.
  Arms: Physical Therapist Group

SUMMARY:
Emergency departments (ED) in several countries integrated physiotherapists in order to reduce wait times for patients with musculoskeletal disorders (MSKD). These initiatives have indeed reduced wait times, length of stay, time waited before seeing a professional and the prescription of unnecessary consultations and diagnostic tests. In Canada, such initiatives are marginal and their effects have not been studied.

The objectives of the project are to evaluate the effects of physiotherapy management of patients with MSKD in ED compared to usual practice on clinical course of patients, use of services and resources, and waiting time and length of stay in ED. The hypothesis is that patients presenting with a MSKD to the ED with direct access to a physiotherapist will have better clinical outcomes and that use of services, waiting time, and length of stay are going to be inferior to those of the EP group.

DETAILED DESCRIPTION:
Background and rationale: Emergency departments (ED) in several countries integrated physiotherapists, which led, for patients with musculoskeletal disorders (MSKD), to a reduction in wait times, length of stay, time waited before seeing a professional and the prescription of unnecessary consultations and diagnostic tests. Furthermore, early access to physiotherapy is associated with a decrease in pain and psychological symptoms and decreased risks of developing persistent pain. In Canada, such initiatives are still marginal and their effects have not been studied.

Objectives: Evaluate the effects of direct access physiotherapy management of patients with MSKD in the ED compared to the usual management by the emergency physician on clinical course of patients (pain, quality of life and disability) and use of services and resources at one and three months, and waiting time and length of stay in the ED.

Methods: A randomized controlled trial is currently in progress at the Centre hospitalier de l'Université Laval (CHUL). Two groups of 50 participants each are recruited over a six months period: one group with direct access to a physiotherapist (PT) in the ED and one control group with the usual access care to the emergency physician. Data is extracted from the patients' medical record, administrative data from the ED, self-administered forms given to the patients during their ED stay and either electronic or phone follow-ups (1 and 3 months). Data will be analysed using descriptive (demographic and clinical profiles) and inferential statistics (repeated ANOVA between groups across time points and Student T tests for independent samples).

Importance of potential findings for MSK health: ED overcrowding causes prolonged lengths of stay, increased rates of patient leaving without being seen, increased medical errors, increased mortality among ambulatory and non-ambulatory patients and decreased patient satisfaction. This project will measure the effects of integrating PTs into the ED in a Canadian hospital setting and help identify ways to improve the current services offered to patients with a MSKD presenting to the ED. Direct access to PT may improve musculoskeletal health outcomes and support positive patient experience.

ELIGIBILITY:
Inclusion Criteria:

* Triage category 3, 4 or 5
* Discharged home with a minor MSKD after ED care
* Able to consent
* Able to understand French and to complete the questionnaire either verbally or in writing

Exclusion Criteria:

* Major MSKD requiring urgent care
* Presence of a red flag or an unstable clinical condition
* Living in a long-term care facility

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2019-06-27 (Actual); Study Completion 2019-06-27 (Actual)

PRIMARY OUTCOMES:
Level of Pain: Numeric Pain Rating Scale | Baseline, 1 and 3 months
  Scale ranging from 0 to 10 where 0 means no pain at all and 10 means the worst pain ever.
Pain Interference on Function: Brief Pain Inventory | Baseline, 1 and 3 months
  List of 10 items (work, sleep, general activity, etc.) represented on a scale ranging from 0 to 10 where 0 means "Does Not Interfere" and 10 means "Completely Interferes". Subscales are averaged and the resulting score is out of 10. A higher score means a higher interference of pain on function.

SECONDARY OUTCOMES:
Pain Catastrophizing: Pain Catastrophizing Scale | Baseline
  List of 13 items (thoughts and feelings about pain) represented on a scale ranging from 0 to 4 where 0 means "Not at all" and 4 means "All the time". Subscales are summed and the resulting score is out of 52. A higher score means a higher tendency to catastrophise pain.
Interventions received by the participants : Standardized Form | Baseline, 1 and 3 months
  Form were every intervention received by the patient was checked as a "Yes" or "No" answer. (Advice, medication, technical aids, referral to another health professional, etc.)
Diagnostic Tests : Standardized Form | Baseline, 1 and 3 months
  Form were every diagnostic test received by the patient was checked as a "Yes" or "No" answer. (X-ray, MRI, CT Scan, ultrasound, etc.)
Consultations with Another Health Professional : Standardized Form | Baseline, 1 and 3 months
  Form were every consultation being prescribed to the patient was checked as a "Yes" or "No" answer.
Satisfaction: Visit-Specific Satisfaction Instrument | Baseline
  List of 7 items (Answers to your questions, Technical skills of the healthcare provider, etc.) represented on a scale ranging from 1 to 5 where 1 means "Excellent" and 5 means "Poor". Subscales are transformed in results out of 100 (1 = 100% and 5 = 0%), averaged and the resulting score is out of 100%. A higher score means higher satisfaction.
Wait Time | Baseline
  Difference between beginning of the intervention and time of arrival between groups during their ED visit
Length of Stay | Baseline
  Difference between departure time and time of arrival between groups during their ED visit

CONTACTS AND LOCATIONS:
Overall Officials: Rose Gagnon, MPT, MSc(c), Principal Investigator — Laval University
Locations (1):
- Centre Hospitalier de l'Université Laval (CHUL), Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gagnon R, Perreault K, Berthelot S, Matifat E, Desmeules F, Achou B, Laroche MC, Van Neste C, Tremblay S, Leblond J, Hebert LJ. Direct-access physiotherapy to help manage patients with musculoskeletal disorders in an emergency department: Results of a randomized controlled trial. Acad Emerg Med. 2021 Aug;28(8):848-858. doi: 10.1111/acem.14237. Epub 2021 Apr 16. PMID 33617696